CLINICAL TRIAL: NCT03336606
Title: Phase Ib Study of a Monoclonal Antibody to OX40 (MEDI0562) Administered Prior to Surgical Resection in Patients With Head and Neck Squamous Cell Carcinoma or Melanoma
Brief Title: Study of MEDI0562 Prior to Surgical Resection in Head and Neck Squamous Cell Carcinoma (HNSCC) or Melanoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Providence Cancer Center, Earle A. Chiles Research Institute (Other); MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017000254
Record Dates: First submitted 2017-10-24; First posted 2017-11-08 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Melanoma; Cell Cancer, Squamous; Carcinoma, Squamous Cell
Keywords: immunotherapy; OX40; antibodies; HNSCC; melanoma; phase 1; squamous cell
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Melanoma; Neoplasms, Squamous Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Intervention Model Description: Patients will be stratified by tumor type and randomly assigned to a MEDI0562 administration schedule; initially 5 patients will enroll to each of two cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (Active Comparator): MEDI0562 administration (90mg on day 1) followed by surgical resection (day 15)
  Interventions: Drug: MEDI0562
- Cohort II (Active Comparator): MEDI0562 administration (30mg on days 1, 3, 5) followed by surgical resection (day 15)
  Interventions: Drug: MEDI0562

INTERVENTIONS:
Drug: MEDI0562 — Surgical resection of tumor
  Other Names: Surgical Resection

SUMMARY:
This clinical trial will evaluate the safety and feasibility of a humanized OX40 agonist, MEDI0562, in the pre-operative setting for patients with head and neck squamous cell carcinoma or melanoma.

DETAILED DESCRIPTION:
This clinical trial is the first to evaluate the safety and feasibility of a humanized OX40 agonist, MEDI0562, in the pre-operative setting for patients with head and neck squamous cell carcinoma or melanoma.

Patients will be randomly assigned to one of two MEDI0562 administration schedules; initially 5 patients will enroll to each cohort. All patients will have a tumor biopsy before administration of MEDI0562 and surgery will be performed on approximately day 15 (+/- 2 days).

There will be a comparison of a surgical specimen to the original biopsy focusing on the composition and immunologic phenotypes of lymphocyte subsets. Although the primary endpoint of this study is immunological, valuable exploratory data on clinical outcomes will also be obtained.

Both the HNSCC and the melanoma patients to be enrolled on this trial are anticipated to have a 50 - 90% probability of recurrence within 5 years after surgery, even with current state-of-the-art post-surgical adjuvant radiation, chemotherapy, or immunotherapy. A recurrence of 25% or less within the 12 months after surgery will be deemed of clinical interest and would inform the design of a larger follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced head and neck squamous cell carcinoma (HNSCC) or stage IIIb/IIIC melanoma who are candidates for R0 surgical resection
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Age 18 years or above
* Laboratory values:

  * WBC ≥2000/uL
  * Hgb >8g/dl (patients may be transfused to reach this level)
  * Platelets >75,000 cells/mm3
  * Serum creatinine 3 X upper limit of laboratory normal
  * Negative bHCG (urine/serum) [women of childbearing potential only]
  * AST (SGOT) and ALT (SGPT) <2.5 X upper limit of laboratory normal
  * Alkaline phosphatase <2.5 X upper limit of laboratory normal
  * Total bilirubin <1.5 X upper limit of laboratory normal, unless due to Gilbert's disease
* INR <1.5, PT <16 seconds, PTT < 38 seconds
* Ability to give informed consent and comply with the protocol
* Anticipated lifespan >12 weeks
* Women of childbearing potential: negative serum/urine pregnancy test <96 hours prior to start of study
* Males and women of childbearing potential: must agree to take appropriate precautions to avoid pregnancy during treatment and through 90 days after last dose of IP

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca/MedImmune staff and/or staff at the study site)
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Receipt of any investigational anticancer therapy during the last 28 days or 5 half-lives, whichever is shorter, prior to the first dose of study treatment
* Any concurrent chemotherapy, investigational agent, biologic, or hormonal therapy for cancer treatment -- concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Local treatment of isolated lesions for palliative intent is acceptable (e.g., local surgery or radiotherapy). -Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug. Note: Local treatment of isolated lesions, excluding target lesions, for palliative intent is acceptable. -Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable. -History of allogenic organ transplantation.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, unstable cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs, or compromise the ability of the patient to give written informed consent -History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥1.5 years before the first dose of investigational product and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease -History of leptomeningeal carcinomatosis -Untreated central nervous system (CNS) metastases and/or carcinomatous meningitis. Note: patients whose brain metastases have been treated may participate provided they show radiographic stability (imaging at least four weeks apart showing no evidence of intracranial progression). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either without the use of steroids or are stable on a steroid dose of ≤10mg/day of prednisone or its equivalent and anti-seizure medications for at least 14 days prior to the start of treatment. Patients on a stable dose of seizure medicines for epilepsy unrelated to cancer are eligible for the trial.
* Active or recent history of diverticulitis. Note: Patients with known diverticulosis are permitted to enroll.
* History of active primary immunodeficiency. -Active infection, including tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and TB testing in line with local practice); hepatitis B (known positive HBV surface antigen (HBsAg) result); hepatitis C; or human immunodeficiency virus (positive HIV 1/2 antibodies). Note: patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Patients with treated HIV, as evidenced by stable CD4 > 200 for at least 6 months, are eligible. -Current or prior use of immunosuppressive medication within 14 days before the first dose of study drug. The following are exceptions to this criterion: • Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)

  • Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease]; diverticulitis [with the exception of diverticulosis]; systemic lupus erythematosus; Sarcoidosis syndrome; or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia • Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement • Any chronic skin condition that does not require systemic therapy • Patients without active disease in the last 5 years may be included but only after consultation with the study physician • Patients with celiac disease controlled by diet alone -Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP -Known allergy or hypersensitivity to study drug(s) or compounds of similar biologic composition to the study drug(s), or any of the study drug excipients. -Any unresolved NCI CTCAE Grade ≥2 toxicities from prior anti-cancer therapy with the exception of vitiligo, alopecia, and the laboratory values defined in the inclusion criteria. -Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician. -Patients with irreversible toxicity not reasonably expected to be exacerbated by study treatment may be included only after consultation with the Study Physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-07-25 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Activation of immune response | 28 days
  The primary objective of this phase Ib clinical trial is to ascertain if there is a difference in immune activation comparing a single dose of MEDI0562 with the equivalent dose divided into a Monday, Wednesday Friday schedule in patients with advanced HNSCC or melanoma. Immune activation will be assessed as a cumulative suppressive index (CSI).

SECONDARY OUTCOMES:
Cancer-related clinical outcomes (progression free survival) | 5 years
  Cancer-related clinical outcomes in patients receiving MEDI0562 will be compared with historical controls for progression free survival.
Cancer-related clinical outcomes (overall survival) | 5 years
  Cancer-related clinical outcomes in patients receiving MEDI0562 will be compared with historical controls for overall survival.
Incidence of Treatment-Emergent Adverse Events in patients with HNSCC or melanoma treated with MEDI0562 (Safety & Tolerability) | 5 years
  The safety of MEDI0562 administration in patients with locally advanced HNSCC and melanoma will be monitored using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Surgical complications after MEDI0562 | 28 days
  Surgical complications after MEDI0562 administration will be monitored using the Clavien-Dindo grading system.

CONTACTS AND LOCATIONS:
Overall Officials: Brenden Curti, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Providence Cancer Center — http://oregon.providence.org/our-services/p/providence-cancer-center/